CLINICAL TRIAL: NCT00002126
Title: A Randomized, Controlled, Multicenter Trial of Filgrastim (Recombinant-Methionyl Human Granulocyte Colony Stimulating Factor; G-CSF) for the Prevention of Grade 4 Neutropenia in Patients With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 087A; GCSF-930101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections; Cytopenias
Keywords: Neutropenia; Granulocyte Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Cytopenia; Neutropenia; Acquired Immunodeficiency Syndrome | interventions — Filgrastim

INTERVENTIONS:
Drug: Filgrastim

SUMMARY:
To determine, in HIV-infected patients, the efficacy of filgrastim ( recombinant-methionyl human granulocyte-colony stimulating factor; G-CSF ) in preventing grade 4 neutropenia, i.e., absolute neutrophil count (ANC) < 500 cells/mm3.

DETAILED DESCRIPTION:
Patients are randomized to receive subcutaneous G-CSF at one of two different doses or no G-CSF (observation) for 24 weeks. Patients who experience ANC < 500 cells/mm3 on two consecutive occasions at least 24 hours apart prior to completing the 24-week study period will be considered to have reached the primary study endpoint; those in the observation group who reach the primary endpoint prior to week 24 may begin receiving G-CSF for the remainder of the study period. After 24 weeks, patients may continue G-CSF on a compassionate basis at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral agents (e.g., AZT, ganciclovir, ddI, ddC), trimethoprim-sulfamethoxazole (Bactrim), interferon, and amphotericin B ONLY IF patient is on the same dose for at least 14 days prior to study entry (patients may not start or stop these agents within 14 days prior to study entry).

Patients must have:

* Documented HIV infection OR history of AIDS.
* CD4 count < 200 cells/mm3.
* ANC (segmental neutrophils plus bands) >= 750 and < 1000 cells/mm3 within 7 days prior to study entry.
* Life expectancy of at least 6 months.

NOTE:

* Stable Kaposi's sarcoma is permitted provided patient does not require myelosuppressive therapy (other than interferon) within 4 weeks prior to study entry.

Prior Medication:

Allowed:

* Prior antiretroviral agents (e.g., AZT, ganciclovir, ddI, ddC), trimethoprim-sulfamethoxazole (Bactrim), interferon, and amphotericin B.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy other than Kaposi's sarcoma and localized basal or squamous cell carcinoma.
* Psychiatric, addictive, or other disorder that compromises ability to give informed consent.
* Known hypersensitivity to E. coli-derived products.

Prior Medication:

Excluded:

* G-CSF, other hematopoietic growth factors (except for erythropoietin), or investigational agents within 14 days prior to study entry.

Substance abuse that would compromise compliance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250

CONTACTS AND LOCATIONS:
Locations (22):
- United States (16):
  - Univ of Alabama at Birmingham / AIDS Outpatient Clinic, Birmingham, Alabama
  - Maricopa County Med Ctr, Phoenix, Arizona
  - CARE Ctr / UCLA Med Ctr, Los Angeles, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Univ Hosp / Univ of Colorado Health Sci Ctr, Denver, Colorado
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Tulane Univ Med School, New Orleans, Louisiana
  - New England Deaconess Hosp, Boston, Massachusetts
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Nalle Clinic, Charlotte, North Carolina
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Kaiser Permanente Med Ctr, Portland, Oregon
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
- Canada (6):
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Toronto Gen Hosp, Toronto, Ontario
  - Wellesley Hosp, Toronto, Ontario
  - Hotel - Dieu de Montreal, Montreal, Quebec
  - Saint Michael's Hosp, Toronto